CLINICAL TRIAL: NCT02795559
Title: Role of Colonic Short Chain Fatty Acids in Obesity: Acute Effects of Inulin and Resistant Starch on Postprandial Short Chain Fatty Acid, Glucose, Insulin, Free-fatty Acid and Gut Hormone Responses
Brief Title: Acute Effects of Dietary Fiber on Postprandial Responses in Lean and Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol Reference # 27112
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Obesity; Diabetes
Keywords: Nutrition; Humans; Obesity; Blood glucose; Dietary fiber; Appetite; Short chain fatty acids
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Glucose; Inulin; Resistant Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean (Other): Subjects within the range of desirable body weight (BMI<25)
  Interventions: Other: Glucose; Other: Inulin; Other: Resistant starch
- OWO (Other): Subjects who are overweight or obese (BMI between 25 and 40)
  Interventions: Other: Glucose; Other: Inulin; Other: Resistant starch

INTERVENTIONS:
Other: Glucose — 75g glucose dissolved in 300ml water
Other: Inulin — 75g glucose plus 24g inulin dissolved in 300ml water
Other: Resistant starch — 75g glucose plus 28g resistant starch in 300ml water

SUMMARY:
It has been suggested that obesity occurs because the colonic microbes in obese individuals, compared to those who are lean, produce more short chain fatty acids during the fermentation of dietary fiber; this means that obese individuals obtain more energy from dietary fiber than lean. On the other hand, it is possible that the ability of colonic short chain fatty acids to improve glycemic control and suppress appetite may be reduced in obese subjects. The aim of this study was to determine the acute effects of 2 fibers commonly used as food ingredients, inulin and resistant starch, on postprandial serum responses of short chain fatty acids, glucose, insulin, free-fatty acids and selected gut hormones in lean and overweight or obese subjects.

DETAILED DESCRIPTION:
The human colon (large intestine) contains hundreds of species of bacteria which exist in a symbiotic (mutually beneficial) relationship with their human host. The number and type of colonic bacteria varies in different people. Recent studies show that overweight individuals have different types of bacteria in their colons than lean subjects, and that as overweight subjects lose weight their colonic bacteria change to resemble those in lean subjects. It was suggested that this was because the bacteria in overweight people more efficiently ferment dietary fiber thus producing more SCFAs and providing more energy to the body. However, this is not consistent with other studies showing that high fiber intakes are associated with reduced risk of obesity.

Some studies have shown that overweight people have higher concentrations of SCFA in their stool samples. But the reasons for the difference in stool concentrations of SCFA have not been studied. Stool concentrations of SCFA may differ in lean and overweight people because of differences in type of bacteria in their colons, differences in dietary intakes or maybe because lean and overweight people absorb SCFA produced by bacteria differently.

Therefore, the objectives of this study were to:

1. determine the relationship between SCFA production and the acute effects of consuming an unabsorbed carbohydrate on blood SCFA, FFA, glucose, insulin, c-peptide and gut hormone responses in lean and overweight subjects
2. determine the types of bacteria in the stools of lean and overweight subjects
3. to see if the types of bacteria are correlated with body weight, the composition of the diet, breath gases, fecal SCFA and other demographic and lifestyle factors.

Healthy subjects with a BMI <25 (lean) or between 25 and 35 (overweight or obese; OWO) took part in a 2 phase study. In phase 1 subjects recorded their dietary intake for 3 days and then provided a stool sample for analysis of micro-organisms and short chain fatty acids. In phase 2 overnight fasted subjects were studied on 3 occasions separated by about a week. On each occasion subjects consumed a control test meal of dextrose, or dextrose plus inulin or dextrose plus resistant start and had breath and blood samples taken at intervals over 4 hours. Subjects were then given a standardized lunch and had more blood and breath samples taken over the next 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age

Exclusion Criteria:

* Pregnant
* BMI<18 or >39.9
* diabetes
* anaemia
* use of diuretics of beta-blockers
* regular user of antibiotics (≥1 course per year over the last 5 years)
* any use of antibiotics within 3 months
* use of laxatives, weight reducing agents, pre/probiotics or supplements known to influence gastrointestinal function within 3 months
* presence of inflammatory bowel disease, malabsorption, motility disorder, gastrointestinal infection, short bowel, or other condition affecting gastrointestinal function
* liver or kidney disease or major medical or surgical event (within the last 6 months) requiring hospitalization
* high fibre intake (>30g/day) or other abnormal dietary pattern
* on a weight-loss diet or not on their habitual diet in the two months prior to the study
* unwilling or unable to give informed consent and/or comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Serum acetate response | 0 to 6 hours after the intervention
  Incremental area under the curve of the serum acetate response from the lowest concentration achieved during the first 3 hours to the end of the study (6hr)

SECONDARY OUTCOMES:
Serum propionate response | 0 to 6 hours after the intervention
  Incremental area under the curve of the serum propionate response from the lowest concentration achieved during the first 3 hours to the end of the study (6hr)
Serum butyrate response | 0 to 6 hours after the intervention
  Incremental area under the curve of the serum butyrate response from the lowest concentration achieved during the first 3 hours to the end of the study (6hr)
Breath hydrogen response | 0 to 6 hours after the intervention
  Incremental area under the curve of the breath hydrogen response from the lowest concentration achieved during the first 3 hours to the end of the study (6hr)
Energy intake | 3 days
  From 3-day diet record, mean energy intake.
Fat intake | 3 days
  From 3-day diet record, mean total fat intake.
Protein intake | 3 days
  From 3-day diet record, mean protein intake.
Carbohydrate intake | 3 days
  From 3-day diet record, mean available carbohydrate intake.
Dietary fiber intake | 3 days
  From 3-day diet record, mean dietary fiber intake.
Fecal microbiota | 1 day
  Ion Torrent V6 16S-rRNA sequencing for comparison of phyla
0-2 hour Glucose response | 0 to 2 hours after consuming treatment
  Incremental area under the curve of the serum glucose response from fasting to 2 hours.
2-4 hour Glucose response | 2 to 4 hours after consuming treatment
  Incremental area under the curve of the serum glucose response from 2 to 4 hours.
Second-meal glucose response | 0 to 2 hours after lunch
  Total area under the curve of the serum glucose response for 2 hours after lunch.
0-2 hour Insulin response | 0 to 2 hours after consuming treatment
  Incremental area under the curve of the serum insulin response from fasting to 2 hours
2-4 hour Insulin response | 2-4 hours after consuming treatment
  Incremental area under the curve of the serum insulin response from 2 to 4 hours.
Second-meal Insulin response | 0-to 2 hours after lunch
  Total area under the curve of the serum insulin response for 2 hours after lunch.
0-2 hour c-peptide response | 0 to 2 hours after consuming treatment
  Incremental area under the curve of the serum c-peptide response from fasting to 2 hours.
2-4 hour c-peptide response | 2 to 4 hours after consuming treatment
  Incremental area under the curve of the serum c-peptide response from 2 to 4 hours.
Second-meal c-peptide response | 0-2 hours after lunch
  Total area under the curve of the serum c-peptide response for 2 hours after lunch.
Free-fatty acid rebound | 0 to 4 hours after consuming intervention
  Increase in serum free-fatty acid concentration from the lowest to the subsequent highest concentration before consuming lunch
Acute total glucagon-like peptide-1 response | 0 to 4 hours after consuming intervention
  Incremental area under the curve of the serum total glucagon-like peptide-1 response from 0 to 4 hours.
Post-lunch total glucagon-like peptide-1 response | 0 to 2 hours after consuming lunch
  Incremental area under the curve of the serum total glucagon-like peptide-1 response from 0 to 2 hours after lunch.
Acute active glucagon-like peptide-1 response | 0 to 4 hours after consuming intervention
  Incremental area under the curve of the serum active glucagon-like peptide-1 response from 0 to 4 hours.
Post-lunch active glucagon-like peptide-1 response | 0 to 2 hours after consuming lunch
  Incremental area under the curve of the serum active glucagon-like peptide-1 response from 0 to 2 hours after lunch.
Acute peptide tyrosine tyrosine response | 0 to 4 hours after consuming intervention
  Incremental area under the curve of the serum PYY response from 0 to 4 hours.
Post-lunch peptide tyrosine tyrosine response | 0 to 2 hours after consuming lunch
  Incremental area under the curve of the serum PYY response from 0 to 2 hours after lunch.
Acute ghrelin response | 0 to 4 hours after consuming intervention
  Incremental area under the curve of the serum ghrelin response from 0 to 4 hours.
Post-lunch ghrelin response | 0 to 2 hours after consuming lunch
  Incremental area under the curve of the serum ghrelin response from 0 to 2 hours after lunch.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No